CLINICAL TRIAL: NCT01758614
Title: The Carotid and Middle Cerebral Artery Occlusion Surgery Study
Acronym: CMOSS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XW125-S001
Record Dates: First submitted 2012-12-24; First posted 2013-01-01 (Estimated); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Carotid Artery Occlusion; Middle Cerebral Artery Occlusion; Stroke
Keywords: carotid artery occlusion; middle cerebral artery occlusion; EC-IC bypass surgery; stroke
MeSH Terms: conditions — Infarction, Middle Cerebral Artery; Stroke | interventions — Coronary Artery Bypass; Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bypass group (Experimental): all the participants in this group will be performed EC-IC bypass surgery
  Interventions: Procedure: bypass surgery
- medical group (Active Comparator): all the participants in this group will be given medical therapy including aspirin 100mg per day or clopidogrel 75mg per day
  Interventions: Drug: Aspirin; Drug: Clopidogrel

INTERVENTIONS:
Procedure: bypass surgery — all participants in this group will be performed EC-IC bypass surgery
  Other Names: EC-IC bypass surgery
  Arms: bypass group
Drug: Aspirin — all participants in this group will be given medical therapy including Aspirin 100mg per day or clopidogrel 75mg per day
  Other Names: Aspirin 100mg per day or clopidogrel 75mg per day
  Arms: medical group
Drug: Clopidogrel
  Arms: medical group

SUMMARY:
The recently published Carotid Occlusion Surgery Study (COSS) failed to show a benefit of extracranial-intracranial (EC-IC) bypass surgery over medical therapy in patients with symptomatic hemodynamically significant carotid occlusion. Since then on, different controversies have been raised on several aspects including the study population, qualifications of surgeons and hemodynamic evaluation.

In COSS protocol, the primary inclusion population is the patient demonstrating occlusion of unilateral ICA while the contralateral ICA less than 50% stenosis. Because of the enrollment problems, in the final result report, 18% patients suffered from contralateral ICA stenosis more than 50%. As we known, COSS utilized oxygen extraction fraction (OEF) ratio by PET as the criterion of hemodynamic evaluation. Bilateral ICAs lesion will disturbed the ratio even the identifying the subgroup of patients with hemodynamic insufficiency.

As an interventional trial, the COSS should ensure the certification for the experienced surgeons. While for expanding the number of centers and enhancing recruitment, COSS made some concessions on the surgeons training and certification. The 15% postoperative event rate is not the best that can be achieved according to recent surgical technical development.

The cerebral hemodynamic insufficiency has been considered as the primary pathophysiological factor for patients with ICA or MCA occlusion. For these patients, antiplatelet therapy is not likely to prevent hemodynamic stroke.EC-IC bypass surgery probably will be the possible effective therapy.

These underlying assumptions deserved further exploration and more strict research.So the CMOSS study in China is designed to compare the efficacy and safety of EC-IC bypass surgery with medical therapy in patients with symptomatic hemodynamically significant carotid occlusion.

DETAILED DESCRIPTION:
Patients with symptoms of cerebral or retinal ischemia associated with ipsilateral internal carotid artery (ICA) occlusion have an annual risk of 5-8% of recurrent ischemic stroke. While in China, the incidence of middle cerebral artery (MCA) occlusion is higher than in western countries. The annual risk of recurrent ischemic stroke in patients with symptomatic ICA or MCA occlusion has not improved over the years. The proportion of recurrence that was minor disabling was rather high.

ELIGIBILITY:
Inclusion Criteria:

* Age ranging between 18 and 65 years;
* Digital subtraction angiography imaging studies demonstrating occlusion of unilateral ICA or MCA;
* Digital subtraction angiography imaging studies demonstrating less than 50% stenosis of any other vessels especially contralateral ICA and MCA;
* Modified Rankin Scales (mRS) 0-2;
* Qualifying TIA or ischemic stroke in the territory of the occluded ICA or MCA must have occurred within the past 12 months;
* The most recent stoke attacked more than 3 weeks ago;
* The neurological deficit must be stable for more than 1 month;
* No massive cerebral infarction (>50% of the MCA territory) in CT or MRI study;
* CT Perfusion demonstrates "misery perfusion" ;
* Competent to give informed consent;
* Legally an adult;
* Geographically accessible and reliable for follow-up;

Exclusion Criteria:

* Other neurovascular disease (such as cerebral aneurysm or arteriovenous malformation) conditions likely to cause focal cerebral ischemia;
* Known unstable angina or myocardial infarction within recent 6 months;
* Pregnant or perinatal stage women;
* Blood coagulation dysfunction;
* Any diseases likely to death within 2 years;
* Past history of EC-IC bypass surgery;
* Any contraindications or allergy to aspirin or clopidogrel;
* Any heart disease likely to cause cerebral ischemia including prosthetic valves, infective endocarditis, atrial fibrillation, sick sinus syndrome, myxoma and cardiomyopathy with ejection fraction less than 25%;
* Allergy to iodine or radiographic contrast media;
* Serum creatinine > 3mg/dl;
* Uncontrolled diabetes mellitus (fasting blood glucose >16.7mmol/l);
* Uncontrolled hypertension (systolic BP >180 mmHg, diastolic BP>110 mmHg);
* Severe liver dysfunction [alanine transaminase (ALT) and/or aspartate aminotransferase (AST) > 3 times of normal level];
* Concurrent participation in any other experimental treatment trial;
* Any condition that in the surgeon's judgment suggests the patient an unsuitable surgical candidate;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2013-06-06 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
the number of participants who suffer from stroke or death after EC-IC bypass surgery or medical therapy | up to 30 days
  The number of participants who suffer from all stroke or death within 30 days after EC-IC bypass surgery or medical therapy
the number of participants who suffer from ipsilateral ischemic stroke | up to 24 months
  the number of participants who suffer from ipsilateral ischemic stroke within 24 months of randomization

SECONDARY OUTCOMES:
the number of participants who suffer from severe transit ischemic attack (TIA) | up to 24 months of randomization
  the number of participants who suffer from severe TIA within 24 months of randomization
the number of participants who suffer from all stroke or death during 30 days to 24 months | during 30 days to 24 months
  the number of participants who suffer from all stroke or death during 30 days to 24 months
the changes from baseline in mRS, national institutes of health stroke scale (NIHSS) and Barthel Index | at 7 days, 30 days, 6 months, 12 months and 24 months
  the changes from baseline in mRS, NIHSS and Barthel Index at 7 days, 30 days, 6 months, 12 months and 24 months
the changes from baseline of cerebral blood flow (CBF) ratio in CT perfusion | at 24 months
  the changes from baseline of CBF ratio in CT perfusion at 24 months
the number of participants who suffer from all kinds of adverse events related to surgery | up to 30 days
  the number of participants who suffer from all kinds of adverse events related to surgery within 30 days in the EC-IC bypass surgery group

CONTACTS AND LOCATIONS:
Overall Officials: Feng Ling, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Department of neurosurgery, Xuanwu hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Powers WJ, Clarke WR, Grubb RL Jr, Videen TO, Adams HP Jr, Derdeyn CP; COSS Investigators. Extracranial-intracranial bypass surgery for stroke prevention in hemodynamic cerebral ischemia: the Carotid Occlusion Surgery Study randomized trial. JAMA. 2011 Nov 9;306(18):1983-92. doi: 10.1001/jama.2011.1610. PMID 22068990
- [Result] Carlson AP, Yonas H, Chang YF, Nemoto EM. Failure of cerebral hemodynamic selection in general or of specific positron emission tomography methodology?: Carotid Occlusion Surgery Study (COSS). Stroke. 2011 Dec;42(12):3637-9. doi: 10.1161/STROKEAHA.111.627745. Epub 2011 Sep 29. PMID 21960571
- [Result] Amin-Hanjani S, Barker FG 2nd, Charbel FT, Connolly ES Jr, Morcos JJ, Thompson BG; Cerebrovascular Section of the American Association of Neurological Surgeons; Congress of Neurological Surgeons. Extracranial-intracranial bypass for stroke-is this the end of the line or a bump in the road? Neurosurgery. 2012 Sep;71(3):557-61. doi: 10.1227/NEU.0b013e3182621488. PMID 22668888
- [Result] Grubb RL Jr, Derdeyn CP, Fritsch SM, Carpenter DA, Yundt KD, Videen TO, Spitznagel EL, Powers WJ. Importance of hemodynamic factors in the prognosis of symptomatic carotid occlusion. JAMA. 1998 Sep 23-30;280(12):1055-60. doi: 10.1001/jama.280.12.1055. PMID 9757852
- [Result] Waaijer A, van der Schaaf IC, Velthuis BK, Quist M, van Osch MJ, Vonken EP, van Leeuwen MS, Prokop M. Reproducibility of quantitative CT brain perfusion measurements in patients with symptomatic unilateral carotid artery stenosis. AJNR Am J Neuroradiol. 2007 May;28(5):927-32. PMID 17494672
- [Derived] Wang T, Yang Y, Wang H, Liu D, Wang J, Luo J, Yang R, Li T, Gong H, Sun X, Derdeyn CP, Ma Y, Jiao L; CMOSS Investigators. CT Perfusion for Predicting Ischemic Stroke in Patients With Symptomatic Carotid or Middle Cerebral Artery Occlusion: A Post Hoc Analysis of the CMOSS Study. Stroke. 2025 Sep;56(9):2579-2587. doi: 10.1161/STROKEAHA.125.051352. Epub 2025 Jun 19. PMID 40534574
- [Derived] Li X, Li Y, Wang T, Sun X, Lu G, Xu X, Yang R, Luo J, Bai X, Tong X, Gu Y, Wang J, Tong Z, Wang Y, Cai Y, Ren J, Wang D, Duan L, Maimaitili A, Hang C, Yu J, Chen T, Ma Y, Jiao L; CMOSS Investigators. Determining the Optimal Age for Extracranial-Intracranial Bypass Surgery: A Post Hoc Analysis of the CMOSS Randomized Trial. Stroke. 2025 Feb;56(2):362-370. doi: 10.1161/STROKEAHA.124.048766. Epub 2024 Dec 27. PMID 39727027
- [Derived] Lu G, Wang T, Sun X, Yang R, Luo J, Tong X, Gu Y, Wang J, Tong Z, Kuai D, Cai Y, Ren J, Wang D, Duan L, Maimaitili A, Hang C, Yu J, Ma Y, Liu S, Jiao L; for CMOSS investigators. Qualifying Event and Recurrence of Ischemic Stroke in Symptomatic Artery Occlusion: A Post Hoc Analysis of CMOSS. J Am Heart Assoc. 2024 Jul 2;13(13):e034056. doi: 10.1161/JAHA.123.034056. Epub 2024 Jun 27. PMID 38934799
- [Derived] Ma Y, Wang T, Wang H, Amin-Hanjani S, Tong X, Wang J, Tong Z, Kuai D, Cai Y, Ren J, Wang D, Duan L, Maimaitili A, Hang C, Yu J, Bai X, Powers WJ, Derdeyn CP, Wu Y, Ling F, Gu Y, Jiao L; CMOSS Investigators. Extracranial-Intracranial Bypass and Risk of Stroke and Death in Patients With Symptomatic Artery Occlusion: The CMOSS Randomized Clinical Trial. JAMA. 2023 Aug 22;330(8):704-714. doi: 10.1001/jama.2023.13390. PMID 37606672
- [Derived] Ma Y, Gu Y, Tong X, Wang J, Kuai D, Wang D, Ren J, Duan L, Maimaiti A, Cai Y, Huang Y, Wang X, Cao Y, You C, Yu J, Jiao L, Ling F. The Carotid and Middle cerebral artery Occlusion Surgery Study (CMOSS): a study protocol for a randomised controlled trial. Trials. 2016 Nov 16;17(1):544. doi: 10.1186/s13063-016-1600-1. PMID 27852286